CLINICAL TRIAL: NCT02104700
Title: Switch From Nevirapine-based Regimen to Once a Day Rilpivirine/Emtricitabine/Tenofovir in Virologically-suppressed HIV-infected Rwandans (Near-Rwanda)"
Brief Title: Switch From Nevirapine-based Regimen to Once a Day Rilpivirine/Emtricitabine/Tenofovir
Acronym: Near-Rwanda
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Philip Grant (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Philip Grant, Associatge Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Near Rwanda; ISR-In-US-264-0123 (Other: Gilead Sciences)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — Rilpivirine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine, Rilpivirine, Tenofovir Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rilpivirine/Emtricitabine/Tenofovir (Active Comparator): "Immediate switch": RILPIVIRINE/ EMTRICITABINE /TENOFOVIR FDC QDAY at randomization.
  Interventions: Drug: Rilpivirine/Emtricitabine/Tenofovir
- Nevirapine/Lamivudine/ plus other NNRTI (Active Comparator): "Delayed switch": Continue NEVIRAPINE 200MG BID + LAMIVUDINE 300MG + OTHER NUCLEOSIDE REVERSE TRANSCRIPTASE INHIBITOR (NRTI) through 24 weeks then switch to RILPIVIRINE 25MG/ EMTRICITABINE 200MG/TENOFOVIR 300MG FDC QDAY and then follow through 48 weeks.
  Interventions: Drug: Rilpivirine/Emtricitabine/Tenofovir

INTERVENTIONS:
Drug: Rilpivirine/Emtricitabine/Tenofovir — Rilpivirine 25mg/Emtricitiabine 200mg/Tenofovir 300mg FDC qday
  Other Names: Complera

SUMMARY:
The study will be an open-label, pilot study in virologically suppressed patients comparing the efficacy, safety and tolerability of two Antiretroviral regimen strategies:

Arm A: "Immediate switch" Rilpivirine/Emtricitabine/Tenofovir (single tablet formulation (STF))at randomization

Arm B: "Delayed switch" Continue Nevirapine/Lamivudine/other Nucleoside reverse transcriptase inhibitor (NRTI)through 24 weeks then switch to STF of Rilpivirine/emtrictabine/tenofovir and followed through 48 weeks.

DETAILED DESCRIPTION:
The current study is designed to be the first study to compare a continued nevirapine-based regimen to a switch to the FDC of rilpivirine/emtricitabine/tenofovir. Rwanda is a model country for implementation of newer approaches to more innovative ART strategies with an excellent National HIV Treatment program in place but has limited experience with clinical trials and as with most African countries has no clinical experience with Rilpivirine in treating HIV infected adults. Done in collaboration with Rwanda Biomedical center.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. A second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test or a previous detectable HIV RNA level
* HIV RNA level below the limit of quantification of the viral load assay in use in-country within the last 12 months
* Screening HIV RNA level below the limit of quantification as defined by the local assay
* At least twelve months of stable first-line antiretroviral therapy consisting of nevirapine and 2 nRTIs approved by the Rwandan HIV Treatment guidelines. (No prior changes in ART are allowed)
* Enrolled in the Rwanda National ART Program with no in-country transfer within the program.
* Negative TB symptom screen or eligible based on algorithm outlined in
* Laboratory values obtained within 30 days prior to study entry:

  * Hemoglobin greater than 8.0 g/dL
  * Platelet count greater than 40,000/mm3
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase less than 5 X ULN
  * Total bilirubin less than 2.5 x ULN
  * Calculated creatinine clearance greater than 60 mL/min as estimated by the Cockcroft-Gault equation:

    * Ability to meet the nutritional requirements for rilpivirine; largest meal should consist of at least 400 total kcals and 117 kcals of fat (13 grams) to be assessed at screening.
    * For women of reproductive potential, negative serum or urine pregnancy test within 4 weeks of initiating study medications and a negative urine pregnancy test at the entry visit prior to randomization.
* "Women of reproductive potential" is defined as women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) and have not undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation).
* Age greater than18 years.
* Ability and willingness of subject to give informed consent.

Exclusion Criteria:

* History of on-treatment virologic failure (defined as HIV RNA level greater than 200 copies/mL at or after 6 months of antiretroviral therapy)
* Any change in prior ART.
* Currently breastfeeding.
* Active tuberculosis.
* Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 14 days prior to study entry.
* NOTE: Isolated cutaneous Kaposi's Sarcoma, oral candidiasis, vaginal candidiasis, mucocutaneous herpes simplex, and other non-serious illnesses (as judged by the site investigator) have no restriction.
* Known allergy/sensitivity to study drugs or their formulations.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Requirement for any current medications that are prohibited with any study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Explore Efficacy | 24 weeks
  To compare proportion of subjects successfully maintaining a plasma viral load <200 copies /mL at week 24 in subjects randomized to rilpivirine/emtricitabine/tenofovir vs. in those randomized to initially continue nevirapine-based ART in this pilot study.

SECONDARY OUTCOMES:
HIV RNA levels | 24 weeks
  To compare between arms the probability of having an HIV RNA level <50 and <400 copies/mL at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zolopa, MD, Principal Investigator — Stanford University
Locations (1):
- Rwanda Military Hospital, Kinombe, Rwanda